CLINICAL TRIAL: NCT05935904
Title: The Progression of Metabolic Syndrome Components During Pregnancy, and the Risks for Adverse Pregnancy Outcomes in Jimma Zone, Southwest Ethiopia: A Prospective Cohort Study.
Brief Title: Progression of Metabolic Syndrome Components During Pregnancy
Acronym: MetS_Preg
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Flemish Interuniversity Council (VLIR) (Network); Jimma University (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0563
Record Dates: First submitted 2023-06-16; First posted 2023-07-07 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Syndrome; Pregnant Women; Birth Outcomes; Dietary Habits; Knowledge, Attitudes, Practice
Keywords: Metabolic syndrome; Cohort; Pregnancy; Birth outcomes; Food culture
MeSH Terms: conditions — Metabolic Syndrome; Feeding Behavior; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Biospecimen Retention: Samples Without DNA — Blood will be collected at baseline, 6 months, and 9 months of pregnancy as well as after birth. Samples of blood will be analyzed for lipid profile and fasting blood glucose. Urine samples will be collected at baseline only for Human chorionic gonadotropin (HCG) test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MetS_risk: Pregnant women in their first trimester who have one or more of the following risk factors: abdominal obesity defined as waist circumference ≥ 2 standard deviations (SD) for gestational age in the first half of pregnancy or presentational BMI >30 kg/m2; triglycerides concentration >150 mg/dl; HDL cholesterol concentrations <50 mg/dL; fasting glucose > 105 mg/dL; and blood pressure > 130/85 mm Hg.
  Interventions: Other: Exposure
- MetS_Free: Pregnant women in their first trimester who are free of any MetS component.
  Interventions: Other: Non exposure

INTERVENTIONS:
Other: Exposure — Dietary habits:
  Data collected using food frequency questionnaire
  Risk factors associated with metabolic syndrome:
  Data collected on nutritional status, biochemical indicators and other risk factors associated with metabolic syndrome progression during pregnancy
  Pregnancy outcomes:
  Adverse pregnancy and birth outcomes.
  Other Names: MetS_Risk
  Groups: MetS_risk
Other: Non exposure — Dietary habits:
  Data collected using food frequency questionnaire
  Risk factors associated with metabolic syndrome:
  Data collected on nutritional status, biochemical indicators and other risk factors associated with metabolic syndrome progression during pregnancy
  Pregnancy outcomes:
  Adverse pregnancy and birth outcomes.
  Other Names: MetS_Free
  Groups: MetS_Free

SUMMARY:
The goal of this cohort study is to investigate the underlying risk factors to develop metabolic syndrome (MetS) during pregnancy, and the associations of MetS and its indicators with birth outcomes in southwest Ethiopia. The study population consists of low-risk pregnant ladies in their first antenatal care visit (ANC), from Jimma Medical center.

The main question[s] it aims to answer are:

i) How do MetS components progress during pregnancy, and what are the underlying risk factors? ii) What is the association between MetS components during early- and late pregnancy and adverse pregnancy outcomes? iii) What is the knowledge, attitude and practices of women toward dietary habits, food taboos, and cultural beliefs during pregnancy?

The study population consists of low-risk pregnant ladies in their first trimester (<15 weeks of pregnancy) in their first antenatal care visit (ANC) who will be followed up until one-month postpartum.

Enrolled women will be assessed four times: at enrolment ≤15 weeks of pregnancy, mid-pregnancy (at 24 weeks), and late pregnancy (at 36 weeks), and within two weeks post-partum for:

1. Sociodemographic data
2. Dietary intake
3. Biochemical analyses
4. Maternal anthropometry:
5. Body composition in a subsample.
6. Knowledge, attitudes and practices of dietary practices during pregnancy
7. Pregnancy and birth outcomes: During the final visit, new born babies will be assessed for Apgar score, weight, length, and head circumference. The mother will be examined for general health and mode of delivery.

DETAILED DESCRIPTION:
Current knowledge about MetS in pregnancy is limited, but it is generally accepted that obesity increases the risk of developing gestational diabetes mellitus (GDM) and preeclampsia (PE). Both of these are associated with an increased risk for developing type 2 diabetes mellitus (T2DM) and cardiovascular disease (CVD) in women later in their life. Poor dietary quality, overweight and/or obesity defined by elevated body mass index (BMI ≥25 kg/m2), are the two most common risk factors associated with the development of MetS during pregnancy. MetS is a serious and escalating public health and clinical challenge in the wake of urbanization, surplus energy intake, and sedentary life habits. MetS during pregnancy can result in complications during pregnancy and can affect the birth outcomes resulting in preterm birth (PB) and fetal growth restriction (FGR) escalating the risk for perinatal mortality and morbidity as well as increasing the risk of developing chronic diseases later in life. Identifying early in pregnancy the unfavourable maternal conditions that can predict poor birth outcomes could help their prevention and management and will warrant a close follow-up for these women from long-term complications. Hence the development of context- and population-specific indicators that define the MetS risk in this population is important in the design of interventions that will be targeting the prevention of MetS.

Study objectives: This study aims to investigate the progression of MetS components during pregnancy, and the associations of MetS components with adverse pregnancy outcomes in the mother-infant cohort study southwest Ethiopia.

Primary aim:

To assess the relationship between maternal MetS components and adverse pregnancy outcomes.

Secondary aima:

i) To assess the progression of MetS components during pregnancy, and the underlying risk factors.

ii) To assess the associations between MetS components during early- and late pregnancy and adverse pregnancy outcomes.

iii) To explore knowledge, attitude and practices toward maternal dietary habits, food taboos, and cultural beliefs during pregnancy.

iv) To develop and validate body composition cut-offs for predicting obesity (as a risk factor for MetS) among Ethiopian pregnant women.

Methodology: A prospective maternal-infant cohort study will be conducted at the Jimma Medical Center, southwest Ethiopia.

The study population consists of low-risk pregnant ladies in their first trimester (<15 weeks of pregnancy) in their first antenatal care visit (ANC) who will be followed up until one-month postpartum.

Recruitment will be at one of the following centers including Jimma Medical center, Shenen Gibe General Hospital, Family Guidance Associations (FGA) and two other health centers.

Enrolled women will be assessed four times: at enrolment ≤15 weeks of pregnancy, mid-pregnancy (at 24 weeks), and late pregnancy (at 36 weeks), and within two weeks post-partum.

Statistical analysis will be conducted using STATA. The progression of MetS components during pregnancy will be assessed using the repeated measures ANOVA procedure. Dietary data and physical activities will be tested as the main risk factors. Log binomial regression analyses will be used to examine the risk for each pregnancy outcome with each of the 5 individual components for MetS and as a composite measure (i.e., MetS). The relative risks, adjusted for maternal body mass index (BMI), age, ethnicity, socioeconomic index, physical activity, smoking status, and fetal sex, will be examined.

Additionally, adapted analyses will be used to define the cutoffs of obesity in this population using maternal body composition data (fat mass and fat-free mass)

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy women with (or without) at least one of the 5 individual components of MetS will be enrolled in the study from each selected health institution if they meet all the inclusion criteria.

Inclusion criteria for the exposed group include additionally:

1. Abdominal obesity defined as waist circumference ≥ 2 standard deviations (SD) for gestational age in the first half of pregnancy or presentational BMI >30 kg/m2, OR
2. Raised triglycerides (>1.70 mmol/l [>150 mg/dl]), OR
3. Reduced high-density lipoprotein cholesterol (<1.29 mmol/l [<50 mg/dl]), OR
4. Raised blood pressure (BP) (i.e., systolic BP >130 mm Hg or diastolic BP >85 mm Hg), OR
5. Raised plasma glucose (>5.6 mmol/l).

Exclusion Criteria:

* Pregnant women with chronic hypertension that necessitates medication, diabetes (also under medication), or any severe chronic illness will not be eligible to participate in the study. Women who have HIV and who take antiretroviral therapy (ART) are also not eligible because of the side effect of ART. Additionally, non-consenting women, ≤18 years old, women who are planning to move outside the study area within the study timeframe due to job transfer or study leave, or those who are not willing to adhere to the prospective follow up visits will not be included in the study. Women whose ultrasound confirmed, twin pregnancy, congenital anomaly or fetal death in utero will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women in their first trimester, who are residents of Jimma town and nearby kebeles (the smallest administrative division or municipality) will be contacted at the selected health institutions and asked to participate in the study. Eligible women who provide their consent will be recruited. Participants will be selected based on their exposure to one or more components of MetS or not. Sampling will be done consecutively until the required sample is reached.
Sampling Method: Non-Probability Sample
Enrollment: 526 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Birth weight | Birth weight will be assessed up to 28 weeks after enrollment
  Birth weight (g)
Infant length | Infant length will be assessed up to 28 weeks after enrollment
  Infant length (cm)
Gestational age at birth | It is measured in weeks, from the first day of the woman's last menstrual cycle to the day of birth.
  Gestational age at birth in weeks will be used to define preterm (babies born alive prior to 37 completed weeks of gestation), term birth (birth between 37 and 42 weeks), and post-term (birth after 42 weeks of gestation).
Preeclampsia (PE) | In all participating women up to 28 weeks after enrollment
  Defined as systolic BP >140 mm Hg or diastolic BP >90 mm Hg, or both, on at least 2 occasions at least 4 hours apart after 20 weeks' gestation but before the onset of labour, or postpartum, with either proteinuria (24-hour urinary protein >300 mg or spot urine protein:creatinine ratio >30 mg/mmol creatinine) or any multisystem complication of PE.
Gestational diabetes (GDM) | In all participating women up to 28 weeks after enrollment
  Defined if fasting glucose of >5.1 mmol/l.

SECONDARY OUTCOMES:
Infant head circumference | Infant head circumference will be assessed up to 28 weeks after enrollment
  Infant head circumference (cm)
High triglyceride concentrations | At baseline and through follow-up up to 28 weeks after enrollment
  High triglyceride level [>150 milligrams per deciliter (mg/dL)]
High-density lipoprotein (HDL) cholesterol | At baseline and through follow-up up to 28 weeks after enrollment
  HDL cholesterol concentrations <50 mg/dL
High blood pressure | At baseline and through follow-up up to 28 weeks after enrollment
  Blood pressure > 130/85 mm Hg
High levels of fasting blood sugar | At baseline and through follow-up up to 28 weeks after enrollment
  Fasting glucose > 105 mg/dL
Maternal weight | Maternal weight will be measured at baseline
  Maternal weight (Kg)
Maternal height | Maternal height will be measured at baseline
  Maternal height (cm)
Dietary intake during six months pregnancy | Assessed at 12 weeks and 24 weeks after enrollment
  Prevalence of women with adequate dietary intake during six months pregnancy

OTHER OUTCOMES:
Prevalence of participants with nutrition knowledge | At baseline in all participants
  Knowledge, attitudes and practices of dietary practices during pregnancy: Using a structured questionnaire, the knowledge, attitudes and practices of the women regarding food taboos and cultural norms during pregnancy will be assessed.
Fat-free mass | At baseline in a sub-sample of participants
  Fat-free mass (Kg) will be measured using the BOD POD.

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, MD, MSc. PhD, Principal Investigator — University Ghent
Locations (1):
- Jimma University Medical Center, Jimma, Ethiopia

IPD SHARING:
Plan to Share IPD: No
All the data both from the main and the secondary outcomes will be used in the analyses and shared as necessary.

REFERENCES:
- [Background] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Background] Muche AA, Olayemi OO, Gete YK. Gestational diabetes mellitus increased the risk of adverse neonatal outcomes: A prospective cohort study in Northwest Ethiopia. Midwifery. 2020 Aug;87:102713. doi: 10.1016/j.midw.2020.102713. Epub 2020 May 19. PMID 32447182
- [Background] Vasilevski V, Carolan-Olah M. Food taboos and nutrition-related pregnancy concerns among Ethiopian women. J Clin Nurs. 2016 Oct;25(19-20):3069-75. doi: 10.1111/jocn.13319. Epub 2016 Jul 14. PMID 27411855
- [Background] Berhe AK, Ilesanmi AO, Aimakhu CO, Mulugeta A. Effect of pregnancy induced hypertension on adverse perinatal outcomes in Tigray regional state, Ethiopia: a prospective cohort study. BMC Pregnancy Childbirth. 2019 Dec 31;20(1):7. doi: 10.1186/s12884-019-2708-6. PMID 31892353
- [Background] Chatzi L, Plana E, Pappas A, Alegkakis D, Karakosta P, Daraki V, Vassilaki M, Tsatsanis C, Kafatos A, Koutis A, Kogevinas M. The metabolic syndrome in early pregnancy and risk of gestational diabetes mellitus. Diabetes Metab. 2009 Dec;35(6):490-4. doi: 10.1016/j.diabet.2009.07.003. PMID 19897394
- [Background] Grieger JA, Bianco-Miotto T, Grzeskowiak LE, Leemaqz SY, Poston L, McCowan LM, Kenny LC, Myers JE, Walker JJ, Dekker GA, Roberts CT. Metabolic syndrome in pregnancy and risk for adverse pregnancy outcomes: A prospective cohort of nulliparous women. PLoS Med. 2018 Dec 4;15(12):e1002710. doi: 10.1371/journal.pmed.1002710. eCollection 2018 Dec. PMID 30513077
- [Background] Aldridge E, Pathirana M, Wittwer M, Sierp S, Leemaqz SY, Roberts CT, Dekker GA, Arstall MA. Prevalence of Metabolic Syndrome in Women After Maternal Complications of Pregnancy: An Observational Cohort Analysis. Front Cardiovasc Med. 2022 Mar 14;9:853851. doi: 10.3389/fcvm.2022.853851. eCollection 2022. PMID 35360031